CLINICAL TRIAL: NCT04058405
Title: Statistical Risk Prediction Models for Adverse Maternal and Neonatal Outcomes in Severe Preeclampsia in a Low-resource Setting, Mpilo Central Hospital, Bulawayo, Zimbabwe.
Brief Title: Risk Prediction Models for Adverse Maternal and Neonatal Outcomes in Preeclampsia
Status: Completed | Type: Observational
Sponsor: Mpilo Central Hospital (Other)
Responsible Party: Principal Investigator, Solwayo Ngwenya, Director, Mpilo Central Hospital
Other Study IDs: MpiloCH
Record Dates: First submitted 2019-08-06; First posted 2019-08-15 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Severe Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Observational — Cross-sectional observations
  Other Names: Studying

SUMMARY:
This proposal describes a single centre retrospective cross-sectional study which will address the need to further develop and test statistical risk prediction models for adverse maternal and neonatal outcomes in low-resource settings; this will be the first such research to be carried out in Zimbabwe.

DETAILED DESCRIPTION:
Hypertensive disorders in pregnancy are a leading cause of maternal and perinatal morbidity and mortality, especially in low-resource settings. Identifying mothers and babies at greatest risk of complications would enable intervention to be targeted to those most likely to benefit from them. However, current risk prediction models have a wide range of sensitivity (42-81%) and specificity (87-92%) indicating that improvements are needed. Furthermore, no predictive models have been developed or evaluated in Zimbabwe.

This proposal describes a single centre retrospective cross-sectional study which will address the need to further develop and test statistical risk prediction models for adverse maternal and neonatal outcomes in low-resource settings; this will be the first such research to be carried out in Zimbabwe.

Data will be collected on maternal demographics characteristics, outcome of prior pregnancies, past medical history, symptoms and signs on admission, results of biochemical and haematological investigations. Adverse outcome will be defined as a composite of maternal morbidity and mortality and perinatal morbidity and mortality. Association between variables and outcomes will be explored using multivariable logistic regression.

Critically, new risk prediction models introduced for our clinical setting may reduce avoidable maternal and neonatal morbidity and mortality at local, national, regional and international level.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included in the study if they have a diagnosis of severe preeclampsia.
* Severe preeclampsia will be defined as high blood pressure (systolic blood pressure (SBP) ≥160, diastolic blood pressure(DBP) ≥110mmHg) and or either severe headaches, epigastric pains and deranged biochemical/haematological blood indices.
* Both singleton and twin/higher order pregnancies will be included.

Exclusion Criteria:

-Women with mild or moderate preeclampsia or less than 20 weeks' of gestation and those with epilepsy will be excluded from the study.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cross-sectional all pregnant women with severe preeclampsia
Sampling Method: Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Maternal death | 3 years
  Binary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: SOLWAYO NGWENYA, PhD, FRCOG, Principal Investigator — Mpilo Central Hospital
Locations (1):
- Mpilo Central Hospital, Bulawayo, Matabeleland, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided
Currently the data is under a university